CLINICAL TRIAL: NCT06350773
Title: The Efficacy of Phosphodiesterase Inhibitors in Patients With Group 2 Pulmonary Hypertension
Brief Title: Phosphodiesterase Type 5 Inhibitors in Patients With Group 2 Pulmonary Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Marina Awad, Assistant Lecturer, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/06122022/ Zaher
Record Dates: First submitted 2024-03-19; First posted 2024-04-05 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Group 2 Pulmonary Hypertension
Keywords: PDEI; pulmonary hypertension; pulmonary vascular resistance; right heart catheterization
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tadalafil-receiving arm (Active Comparator): Patients will take tadalafil for the 12 week period of follow up, in addition to the standard evidence-based therapy for the left heart disease.
  Interventions: Drug: tadalafil 20 mg then 40 mg if tolerated
- Tadalafil non-receiving arm (No Intervention): Patients will not take tadalafil for the 12 weeks follow up, only standard evidence-based therapy for the left heart disease.

INTERVENTIONS:
Drug: tadalafil 20 mg then 40 mg if tolerated — Patients will receive tadalafil for 12 week follow up period, in addition to the conventional anti failure therapy.
  Arms: tadalafil-receiving arm

SUMMARY:
The goal of this clinical trial is to test the efficacy of tadalafil in patients with group II pulmonary hypertension with elevated pulmonary vascular resistance (PVR). The main question it aims to answer is:

• Can tadalafil improve patients with group II pulmonary hypertension with elevated PVR? Participants will undergo right heart catheterization (RHC) to make sure they are fulfilling the inclusion criteria, then will be asked to take tadalafil 20 mg for two weeks then 40 mg if tolerated for 12 weeks, then participants will be followed up. Investigators will compare the drug group with another age- and sex- matched control placebo group.

DETAILED DESCRIPTION:
The study aims at studying the efficacy of tadalafil in patients with group 2 pulmonary hypertension with elevated pulmonary vascular resistance guided by RHC. After fulfilling the inclusion criteria, investigators will recruit 48 patients, and do baseline echocardiography for comprehensive right ventricular (RV) study and 6 minute walk test, and then start tadalafil 20 mg then 4mg if tolerated, for 24 patients (drug group). After three months follow up, investigators will follow up the patients regarding RV function and the functional capacity, compared to matched control group.

ELIGIBILITY:
Inclusion Criteria:

* group 2 pulmonary hypertension with precapillary component with PVR more than 4 by RHC
* Patients should be on HF medical therapy 90 days before enrollment in the study.

Exclusion Criteria:

* Anticipated cardiac resynchronization therapy within 3 months of enrollment.
* Hypersensitivity, allergy, or intolerable side effects of PDE-5 inhibitors.
* Contraindication to PDE-5 inhibitors, including current nitrate therapy.
* All groups of PH, other than group 2 PH (isolated post capillary pulmonary hypertension).
* History of heart transplant, ventricular-assist device, or any other solid-organ transplant
* Likely to have solid-organ transplant or any other major surgery during study enrollment/treatment period.
* Female subject who is pregnant, breast-feeding, or unwilling to practice an acceptable method of birth control unless postmenopausal or sterile.
* Unreliability as a study participant, based on the investigator's (or designee's) knowledge of the subject (e.g., alcohol or other substance abuse, inability or unwillingness to adhere to the protocol, documented noncompliance, or vulnerable population)
* Current enrollment, or enrollment completed <30 days previously, in another investigational drug or device clinical study.
* Undergoing dialysis for end-stage renal disease.
* End-stage liver disease comorbidities, limiting exercise tolerance.
* Morbid obesity (body mass index > 40).
* Severe peripheral vascular disease with intermittent claudication.
* Status after amputation of lower extremity(s) at any level.
* Severe degenerative joint disease preventing normal walking.
* Cerebrovascular accident with long-term sequelae affecting ability to walk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Functional capacity of the patients | 12 weeks
  Six minute walk test, to assess the number of meters the patient can walk within 6 minutes, in be measured in meter unit.
heart failure symptoms | 12 weeks
  using NYHA classification either 1, 2, 3 or 4

SECONDARY OUTCOMES:
right ventricular function | 12 weeks
  using Echocardiography, by measuring
  * RV diameters (basal, mid cavity and longitudinal) in mm
  * Transannular plane systolic excursion (TAPSE) in mm.
right ventricular function | 12 weeks
  * Fractional area change (FAC) in percentage.
  * RV strain in percentage.
right ventricular function | 12 weeks
  - Tricuspid regurgitation severity by measuring jet area in cm2.
right ventricular function | 12 weeks
  using Echocardiography, by measuring pulmonary artery systolic pressure in mmHg.
right ventricular function | 12 weeks
  using Echocardiography, by measuring right ventricular systolic and diastolic velocities in cm/sec.

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Ahmed Abdelhady, Doctorate, Study Director — Beni-Suef University
Locations (1):
- Beni Suef University, Cairo, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No